CLINICAL TRIAL: NCT04176783
Title: Carolina's Opioid Reduction Effort
Brief Title: Opioid-Free Orthopaedic Surgery
Acronym: CORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9120
Record Dates: First submitted 2018-04-16; First posted 2019-11-25 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Analgesics, Opioid; Methods; Analgesics, Non-Narcotic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid (Active Comparator): The opioid-based arm utilizes traditional, standard-of-care treatment for each applicable surgery. The medications (including dosage and frequency) used in this arm vary depending on the surgery being performed; however, tend to include medications in the opioid family such as Hydromorphone, Hydrocodone, Tramadol, or Oxycodone.
  Interventions: Drug: Opioids
- Opioid-Free (Active Comparator): The opioid-free arm utilizes medications that do not belong to the opioid family of medications. All medications used are FDA-approved and no experimental medications are being used. The medications (including dosage and frequency) used in this arm vary depending on the surgery being performed; however, tend to include medications such as Gabapentin, Tylenol, Meloxicam, Bupivacaine, or Ketorolac.
  Interventions: Drug: Opioid-Free

INTERVENTIONS:
Drug: Opioids — narcotic pain medicine
  Other Names: Control
  Arms: Opioid
Drug: Opioid-Free — non narcotoc pain medication
  Other Names: Intervention; Non-Opioid
  Arms: Opioid-Free

SUMMARY:
To compare the safety and effectiveness of two pain control pathways following routine orthopaedic surgical procedures (single level or two-level ACDF/ACDA, 1st CMC arthroplasty, Hallux Valgus/Rigidus corrections, diagnostic knee arthroscopies, total hip arthroplasty, and total shoulder arthroplasty / reverse total shoulder arthroplasty). The control group will undergo surgery with an opioid-based pain protocol and the intervention group will undergo surgery with a multimodal, opioid-free protocol.

Patients will have data collected with respect to pain scores, overall comfort level, overall satisfaction with the surgical experience and recovery, constipation, falls, and overall satisfaction with pain control, in addition to procedure-specific outcome scores and patient-specific metrics.

ELIGIBILITY:
Inclusion Criteria

1. Patient is scheduled to undergo one of the following procedures:

* Primary single-level or two-level ACDF or ACDA for degenerative disease
* Primary 1st CMC arthroplasty
* Primary Hallux Valgus or Hallux Rigidus correction
* Diagnostic knee arthroscopy +/- meniscal debridement
* Elective primary total shoulder or reverse total shoulder arthroplasty
* Primary total hip arthroplasty

Exclusion Criteria

1. Revision surgery for one of the study-specific procedures
2. Chronic opioid therapy - per investigator discretion
3. Significant liver disease - (NOTE: Patients with a history of liver disease will have a hepatic panel drawn to be reviewed by the study investigator to asses if the values are within acceptable limits for inclusion in the study)
4. Fracture or soft tissue injury
5. Sickle cell disease
6. Workers compensation
7. Alcohol dependence
8. Contra-indication to regional anesthesia
9. History of gastrointestinal (GI) bleeding or peptic ulcer
10. History of bleeding problems
11. Patients taking anticoagulants, not including aspirin (only applies to Randomized portion of study. These patients can still participate in Observational Control Group)
12. Renal insufficiency - Creatinine clearance less than 30 mL/min (only applies to patients having surgery requiring NSAIDs treatment)
13. Outpatient THA or TSA/RTSA
14. Hammertoe in isolation (Hallux Valgus/Rigidus exclusion only)
15. Concomitant meniscal repair or microfracture (Knee Arthroscopy exclusion only)
16. Ineligible for spinal anesthesia (THA exclusion only)
17. Previous ipsilateral hip surgery, not including hip scope (THA exclusion only)
18. Allergy to non-steroidal anti-inflammatory medications (NSAIDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain at 24 hours postop | 24 hours
  Numeric Pain Rating Scale 0-10, with 10 representing the highest/worst pain score

SECONDARY OUTCOMES:
Pain at 6 hours postop | 6 hours
  Numeric Pain Rating Scale 0-10, with 10 representing the highest/worst pain score
Pain at 12 hours postop | 12 hours
  Numeric Pain Rating Scale 0-10, with 10 representing the highest/worst pain score
Pain at 2 weeks postop | 2 weeks
  Numeric Pain Rating Scale 0-10, with 10 representing the highest/worst pain score
Pain at 6 weeks postop | 6 weeks
  Numeric Pain Rating Scale 0-10, with 10 representing the highest/worst pain score
Pain at 1 year postop | 1 year
  Numeric Pain Rating Scale 0-10, with 10 representing the highest/worst pain score
General Health | 1 year
  Veterans Rand-12

CONTACTS AND LOCATIONS:
Overall Officials: Nady M Hamid, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina, P.A., Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Derived] Shing EZ, Leas D, Michalek C, Wally MK, Hamid N. Study protocol: randomized controlled trial of opioid-free vs. traditional perioperative analgesia in elective orthopedic surgery. BMC Musculoskelet Disord. 2021 Jan 23;22(1):104. doi: 10.1186/s12891-021-03972-9. PMID 33485328